CLINICAL TRIAL: NCT02374697
Title: Assessment of Tele-expertise for Second Medical Opinion on Pathological Diagnosis
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Agence Regionale de Sante d'Ile de France (Other Government)
Responsible Party: Sponsor
Other Study IDs: TLM-Pathology Expertise
Record Dates: First submitted 2015-02-05; First posted 2015-03-02 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-06

CONDITIONS: Anatomical Pathological Condition
Keywords: Second opinion
MeSH Terms: conditions — Pathological Conditions, Anatomical

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fixed tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Before tele-expertise: Usual second opinion with pathological slides sent by mailing
- During Tele-expertise: Second opinion with tele-expertise
  Interventions: Device: During tele-expertise

INTERVENTIONS:
Device: During tele-expertise
  Groups: During Tele-expertise

SUMMARY:
The purpose of this study is to determine whether digitalizing pathological slides and let it accessible on a server for a second medical opinion (tele-expertise) would reduce the time to diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* All patients in need for a second medical opinion on a pathological sample

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in need for a second medical opinion on a pathological sample
Sampling Method: Non-Probability Sample
Enrollment: 470 (Actual)
Dates: Start 2013-09; Primary Completion 2015-06 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Delay of second medical opinion | Up to 10 weeks
  Between preparation of the slide and the result

SECONDARY OUTCOMES:
Number of second medical opinion requested | During the whole study (around 8 months)
Overall costs | Within 6 months after the start of tele-expertise
  Sum of the durations of the professionals immobilization for performing a diagnosis x wages + costs of the telemedicine solution development and implementation.
Number of times that the pathologist who gave the second opinion required the original material | During the whole study (around 8 months)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Guettier, MD, PhD, Principal Investigator — Hôpital Bicêtre. Assistance Publique - Hôpitaux de Paris; Isabelle Durand-Zaleski, MD, PhD, Principal Investigator — DRCD URC Eco. Assistance Publique - Hôpitaux de Paris
Locations (11):
- France (11):
  - Hôpital Saint Antoine, Paris, Paris
  - Centre de Pathologie- Bièvres, Bièvres
  - Hôpital Henri Mondor, Créteil
  - Centre Hospitalier Simone Veil, Eaubonne
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Bichat, Paris
  - Hôpital Cochin, Paris
  - Hôpital Saint Louis, Paris
  - Centre Hospitalier René Dubos, Pontoise
  - Hôpital Paul Brousse, Villejuif
  - Centre Hospitalier de Villeneuve Saint Georges, Villeneuve-Saint-Georges

REFERENCES:
- [Background] Kidholm K, Ekeland AG, Jensen LK, Rasmussen J, Pedersen CD, Bowes A, Flottorp SA, Bech M. A model for assessment of telemedicine applications: mast. Int J Technol Assess Health Care. 2012 Jan;28(1):44-51. doi: 10.1017/S0266462311000638. PMID 22617736
- [Derived] Charrier N, Zarca K, Durand-Zaleski I, Calinaud C; ARS Ile de France telemedicine group. Efficacy and cost effectiveness of telemedicine for improving access to care in the Paris region: study protocols for eight trials. BMC Health Serv Res. 2016 Feb 8;16:45. doi: 10.1186/s12913-016-1281-1. PMID 26857558